CLINICAL TRIAL: NCT00743145
Title: Effects of Low-dose Naltrexone in Combination With a Range of Smoked Marijuana
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Research Foundation for Mental Hygiene, Inc. (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Margaret Haney, Clinical Psychaitrist, New York State Psychiatric Institute
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB# 5693; DA19239 (Other Grant/Funding Number: National Institute on Drug Abuse (NIDA))
Record Dates: First submitted 2008-08-26; First posted 2008-08-28 (Estimated); Results first posted 2018-09-14 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-08

CONDITIONS: Marijuana Smoking
Keywords: naltrexone; smoked marijuana; marijuana use
MeSH Terms: conditions — Marijuana Smoking; Marijuana Use | interventions — Dronabinol; nabiximols; Naltrexone

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind, placebo-controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Placebo naltrexone + Inactive marijuana (Placebo Comparator): Placebo naltrexone capsules (0mg), inactive marijuana (0% THC). Each study participant underwent 8 conditions in a randomized order.
  Interventions: Drug: Inactive Marijuana (0% THC); Drug: Placebo naltrexone
- Placebo naltrexone + Active marijuana (5.5% THC) (Placebo Comparator): Placebo naltrexone capsules (0mg), active marijuana (5.5% THC). Each study participant underwent 8 conditions in a randomized order.
  Interventions: Drug: Active Marijuana (5.5% THC); Drug: Placebo naltrexone
- Placebo naltrexone + Active marijuana (6.2% THC) (Placebo Comparator): Placebo naltrexone capsules (0mg), active marijuana (6.2% THC). Each study participant underwent 8 conditions in a randomized order.
  Interventions: Drug: Active Marijuana (6.2% THC); Drug: Placebo naltrexone
- Naltrexone + Active marijuana (5.5% THC) (Experimental): Naltrexone capsules (12mg), active marijuana (5.5% THC). Each study participant underwent 8 conditions in a randomized order.
  Interventions: Drug: Active Marijuana (5.5% THC); Drug: Naltrexone
- Naltrexone + Active marijuana (6.2% THC) (Experimental): Naltrexone capsules (0mg), active marijuana (6.2% THC). Each study participant underwent 8 conditions in a randomized order.
  Interventions: Drug: Active Marijuana (6.2% THC); Drug: Naltrexone
- Naltrexone + Inactive marijuana (Placebo Comparator): Naltrexone capsules (12mg), inactive marijuana (0% THC). Each study participant underwent 8 conditions in a randomized order.
  Interventions: Drug: Inactive Marijuana (0% THC); Drug: Naltrexone

INTERVENTIONS:
Drug: Inactive Marijuana (0% THC) — Marijuana cigarette containing 0% THC
  Other Names: Cannabis
  Arms: Naltrexone + Inactive marijuana; Placebo naltrexone + Inactive marijuana
Drug: Active Marijuana (5.5% THC) — Marijuana cigarette containing 5.5% THC
  Other Names: Cannabis
  Arms: Naltrexone + Active marijuana (5.5% THC); Placebo naltrexone + Active marijuana (5.5% THC)
Drug: Active Marijuana (6.2% THC) — Marijuana cigarette containing 6.2% THC
  Other Names: Cannabis
  Arms: Naltrexone + Active marijuana (6.2% THC); Placebo naltrexone + Active marijuana (6.2% THC)
Drug: Naltrexone — Naltrexone (12mg/70kg)
  Other Names: Revia
  Arms: Naltrexone + Active marijuana (5.5% THC); Naltrexone + Active marijuana (6.2% THC); Naltrexone + Inactive marijuana
Drug: Placebo naltrexone — Naltrexone (0mg)
  Other Names: PBO
  Arms: Placebo naltrexone + Active marijuana (5.5% THC); Placebo naltrexone + Active marijuana (6.2% THC); Placebo naltrexone + Inactive marijuana

SUMMARY:
In heavy marijuana smokers, opioid receptor blockade increases the subjective and cardiovascular effects of marijuana. The current study was designed to clarify opioid-cannabinoid interactions by assessing how naltrexone shifts the dose-response function for marijuana-elicited effects in heavy marijuana smokers. For this within-subject, double-blind study, a marijuana smoking procedure was designed to characterize a dose-response relationship for marijuana's subjective and cardiovascular effects under blinded conditions.

ELIGIBILITY:
Inclusion Criteria:

* Current marijuana use
* Able to perform study procedures
* Women practicing an effective form of birth control

Exclusion Criteria:

* Current repeated illicit drug use (other than marijuana)
* Presence of significant medical illness (e.g., diabetes, cardiovascular disease,hypertension, hepatitis, clinically significant laboratory abnormalities, LFTs > 3x upper limit of normal, blood pressure > 140/90

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2008-05; Primary Completion 2009-07 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Haney, Ph.D., Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo, Naltrexone, Marijuana: A total of 23 participants enrolled but only 19 completed. All patients participated in all conditions; they were randomized to placebo or naltrexone treatment in a counterbalanced fashion, and underwent all smoking conditions in separate, counterbalanced sessions.
Period: Overall Study
Arm/Group | Placebo, Naltrexone, Marijuana
Started | 23
Completed | 19
Not Completed | 4
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 2
Not completed — Pregnancy | 1

BASELINE CHARACTERISTICS:
Population: 19 participants completed the study.
Groups:
- Placebo, Naltrexone, Marijuana: During each of the 8 outpatient sessions, participants smoked a total of 6 puffs from 3 marijuana cigarettes (2 puffs from each cigarette). Marijuana administration occurred 45 minutes after capsule administration. The number of active versus inactive cigarettes smoked during each session varied, according to active puff conditions (i.e., 0 puffs = 3 inactive cigarettes; 2 puffs = 1 active + 2 inactive cigarette; 4 puffs = 2 active + 1 inactive cigarette; 6 puffs = 3 active + 0 inactive cigarette). Cigarettes were color coded, indicating the order in which they were to be smoked and active cigarettes were always smoked before inactive. A within-subject design was used in which all participants were exposed to each of the puff conditions in combination with naltrexone or placebo. The order of naltrexone dosing and puff condition was randomized within the session and across participants.
Arm/Group | Placebo, Naltrexone, Marijuana
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.0 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 8
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Subjective Marijuana Effects
Description: Subjective ratings of marijuana's quality and effect ('Strength', 'Good Effect', 'High', 'Stimulation') and craving ('Want Marijuana') as a function of active puffs and naltrexone, using a visual analogue scale with a series of 100 mm long lines labeled 'not at all' at one end (0 mm) and 'extremely' at the other end (100 mm). Participants were instructed to indicate how they felt at that particular moment. Higher ratings indicate more agreement with the statement.
Time Frame: 180 minutes after marijuana administration, during each of 8 outpatient sessions over the course of 3-6 weeks.
Measure: Mean (Standard Error); unit: units on a scale (0-100mm)
Arm/Group | Placebo Naltrexone + Inactive Marijuana | Placebo Naltrexone + Active Marijuana (5.5% THC) | Placebo Naltrexone + Active Marijuana (6.2% THC) | Naltrexone + Active Marijuana (5.5% THC) | Naltrexone + Active Marijuana (6.2% THC) | Naltrexone + Inactive Marijuana
Number analyzed (Participants) | 19 | 19 | 19 | 19 | 19 | 19
units on a scale (0-100mm)
  "Marijuana Strength" | 13 (1) | 15 (1) | 16 (2) | 16 (2) | 20 (2) | 16 (2)
  "Marijuana Good Effect" | 14 (2) | 37 (3) | 30 (2.5) | 31 (3) | 46 (2) | 26 (2)
  "Marijuana High" | 10 (1) | 10.5 (0.5) | 10 (1) | 11 (1.5) | 16 (1.5) | 10 (1.5)
  "Marijuana Stimulation" | 16 (2) | 20 (2) | 16 (2) | 20 (1.5) | 30 (2) | 22 (2)
  "Want Marijuana" | 50 (1.5) | 48 (1) | 37 (1.5) | 49 (1) | 45 (1.5) | 50 (1.5)

ADVERSE EVENTS:
Time Frame: 4 weeks for each treatment and 1 week after receiving last treatment.
Description: Safety population included all participants who received at least one intervention. Research staff routinely asked participants to report any adverse events occurring during study sessions and during outpatient washout periods.
Groups:
- Placebo Naltrexone + Inactive Marijuana (0.0% THC): 0mg naltrexone + 0.0% THC marijuana
- Placebo Naltrexone + Active Marijuana (5.5% THC): 0mg naltrexone + 5.5% THC marijuana
- Placebo Naltrexone + Active Marijuana (6.2% THC): 0mg naltrexone + 6.2% THC marijuana
- Naltrexone + Inactive Marijuana (0.0% THC): 12mg naltrexone + 0.0% THC marijuana
- Naltrexone + Active Marijuana (5.5% THC): 12mg naltrexone + 5.5% THC marijuana
- Naltrexone + Active Marijuana (6.2% THC): 12mg naltrexone + 6.2% THC marijuana
Arm/Group | Placebo Naltrexone + Inactive Marijuana (0.0% THC) | Placebo Naltrexone + Active Marijuana (5.5% THC) | Placebo Naltrexone + Active Marijuana (6.2% THC) | Naltrexone + Inactive Marijuana (0.0% THC) | Naltrexone + Active Marijuana (5.5% THC) | Naltrexone + Active Marijuana (6.2% THC)
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23 | 0/23 | 0/23 | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23 | 0/23 | 0/23 | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23 | 0/23 | 0/23 | 0/23 | 0/23

LIMITATIONS AND CAVEATS:
This study is limited by its small sample size, and portion of males to females.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No